CLINICAL TRIAL: NCT02016092
Title: Proteomics, Metabolomics, Lipidomics and Genetic Analysis for Biomarker DISCOVERY in Parkinson's Disease
Brief Title: Biomarker Discovery in Parkinson's Disease
Acronym: DISCOVERY-PD
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: The Parkinson's Institute (Other)
Responsible Party: Principal Investigator, Birgitt Schuele, Associate Professor, The Parkinson's Institute
Other Study IDs: ECH-13-24; 5258 (Other Grant/Funding Number: Berg Pharma, LLC)
Record Dates: First submitted 2013-12-14; First posted 2013-12-19 (Estimated); Last update posted 2016-03-14 (Estimated); Status verified 2016-03

CONDITIONS: Parkinson's Disease
Keywords: Parkinson's disease; biomarkers; blood; urine,; proteomics; lipidomics; metabolomics
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Blood & Urine Specimen Collection: Up to 20mL of venous blood samples will be collected for plasma multi-omic analysis, as well as optional genetic, analyses.
  Urine samples (~50ml) will be collected via sterile urine cup and transferred into appropriate urine tube for multi-omic analysis.
  All Samples may be saved for future studies, if consented.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Patients with Parkinson's disease
- Healthy Controls

SUMMARY:
There are approximately one million Americans who live with Parkinson's disease with 50,000 new cases per year and this rate is expected to rise with an aging population. The underlying pathophysiology and disease understanding of PD still remains elusive due to a combination of disease complexity and lack of predictive capability of existing models.

The Berg Interrogative Biology™ discovery platform has demonstrated a unique capability in producing drug targets and biomarkers that truly represent a disease phenotype. It has been able to catalyze molecules now in late stage clinical trials in cancer and many pre-clinical candidate therapeutics and biomarkers in endocrinology and central nervous system (CNS) diseases. The platform is able to decipher normal versus disease signatures by integration of data sets from the genome, metabolome, proteome, and lipidome in an agnostic manner that is subjected to Bayesian Artificial Intelligence informatics. The resulting nodes are then put back into wet-lab validation before proceeding to proof-of-principle pre-clinical testing.

By utilizing clinical data and specimens obtained by the medical specialists at The Parkinson's Institute, along with Berg's Interrogative Biology™, this study aims to discover a disease biomarker enabling the creation of a diagnostic test for Parkinson's disease.

ELIGIBILITY:
Inclusion Criteria:

For PD cases:

Inclusion Criteria:

* Men and women with the clinical diagnosis of idiopathic PD
* Willing and able to give informed consent
* Willing and able to comply with scheduled visits, required study procedures and laboratory tests

Exclusion Criteria:

PD Subjects with any of the following may not be enrolled:

1. Presence of atypical or secondary parkinsonism
2. Inability to provide a blood and/or urine sample
3. History of renal failure and/or on dialysis
4. Currently taking a medication in the following categories: dopamine blockers, neuroleptics, and/or dopamine blocking agents.
5. Any medical, psychiatric or other condition which, in the opinion of the investigator, would preclude participation

Healthy Controls:

All of the following criteria must be met for a Healthy Control to be enrolled in the study:

1. Healthy controls with no diagnosis of PD and any of the exclusion criteria
2. Willing and able to give informed consent
3. Willing and able to comply with scheduled visits, required study procedures and laboratory tests

Healthy Controls with any of the following may not be enrolled:

1. No clinically significant or unstable medical or psychiatric condition that would interfere with the conduct of the study
2. Diagnosis of PD or presence of signs of a neurodegenerative disorder, e.g. essential tremor
3. First degree relative with PD/parkinsonism
4. Inability to provide a blood and/or urine sample
5. History of renal failure and/or on dialysis
6. Any medical, psychiatric or other condition which, in the opinion of the investigator, would preclude participation

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Parkinson's patients
Sampling Method: Probability Sample
Enrollment: 400 (Actual)
Dates: Start 2013-12; Primary Completion 2016-03 (Actual); Study Completion 2016-06 (Estimated)

PRIMARY OUTCOMES:
Biological markers of Parkinson's disease | 18 months
  To identify biologic markers of Parkinson's Disease (PD) for use in diagnostic testing.

SECONDARY OUTCOMES:
Correlation between biologic markers and clinical features of PD | 36 months
  To identify and investigate possible correlations between biologic markers and clinical features of PD.

CONTACTS AND LOCATIONS:
Locations (1):
- The Parkinson's Institute and Clinical Center, Sunnyvale, California, United States

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be made available, summary datasets may be published in peer-review journals.